CLINICAL TRIAL: NCT05568056
Title: The Efficacy of a Visualizing Reading Intervention on Improving the Brain's Reading Network in Children With Autism
Brief Title: Efficacy of Reading Intervention on the Brain Connectivity in Autism
Acronym: BrainREAD
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 19-03-2120
Record Dates: First submitted 2022-09-27; First posted 2022-10-05 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder; Autism; Reading Problem
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: ASD participants randomly assigned to Experimental or Waitlist control groups. NT-EXP participants assigned to experimental group NT participants assigned to waitlist control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASD-EXP and NT-EXP (Experimental): Autistic children and Neurotypical children who receive intervention between pre and post testing
  Interventions: Behavioral: Visualizing and Verbalizing for Language comprehension and Thinking
- ASD-WLC and NT (No Intervention): Autistic children who receive intervention only after their pre and post testing and Neurotypical children who do not receive any intervention

INTERVENTIONS:
Behavioral: Visualizing and Verbalizing for Language comprehension and Thinking — The V/V intervention program is a language remediation program designed by Dr. Nanci Bell, and developed by the Lindamood-Bell Learning Processes (LBLP) (Bell, 1991b). It has been widely used among children with reading disorders, but not with children with ASD. This intervention is based on the use of nonverbal sensory input, in the form of imaged gestalts, in order to develop oral and written language comprehension, establish vocabulary, and develop higher order thinking skills (Bell, 1991a,b).
  Arms: ASD-EXP and NT-EXP

SUMMARY:
The overarching goal of this proposal is to test the impact of a comprehensive reading intervention program (Visualizing and Verbalizing) on changing the neurobiological mechanisms underlying reading comprehension deficits in children with autism spectrum disorders (ASD). To this end, the investigators will test a group of children with ASD and NT control participants who share common characteristic of average level decoding along with below average reading comprehension. Inclusion of an additional NT group that does not have any reading comprehension deficit will provide another control for additional comparisons.

DETAILED DESCRIPTION:
The overarching goal of this proposal is to test the impact of a comprehensive reading intervention program on changing the neurobiological mechanisms underlying reading comprehension deficits in children with autism spectrum disorders (ASD). There is evidence that as many as 65% of children with ASD have a deficit in reading comprehension. This ultimately has profound impact on language, learning, and academic success (Nation, Clarke, Wright, & Williams, 2006). Poor reading comprehension in children with autism is often masked by their relative strength in decoding. Moreover, reading comprehension in general is not well-understood, and as a result, current treatments are limited in its potential and in its effectiveness. In this project, the investigators will test a group of children with ASD and NT control participants who share common characteristic of average level decoding along with below average reading comprehension. The investigators also have included an additional NT group without any reading comprehension deficits, and this group will serve as another control for additional comparisons. The investigators will test the efficacy of an intensive reading intervention training program, visualizing and verbalizing for language comprehension and thinking (V/V), and its effects on changing the brain circuitry underlying reading comprehension in children with ASD. The project will use multimodal neuroimaging with task-based functional MRI, resting state functional MRI, diffusion imaging, and neuropsychological testing. It should be noted that neuroimaging as well as behavioral studies of language in autism have largely ignored a subgroup of children with comprehension deficits. The proposed project addresses this critical gap by targeting brain plasticity in children with ASD (age: 7-13 years). Average decoding ability with below average comprehension of language in children is an important problem of academic and public health significance. The outcome of this study will throw more light on this important subgroup of children. In addition, it will test the efficacy of an intervention that can, in the long-run, help NT and children with reading problems to achieve academic success. Findings may provide important preliminary steps in using V/V intervention in schools.

This project will use multimodal neuroimaging [functional MRI, structural MRI, and diffusion weighted imaging (DWI)] to assess changes in brain function and white matter connectivity in autism. This will be accomplished using 4 groups of participants matched on age, gender and IQ: 1) children with ASD who will undergo the V/V intervention after their first MRI scan (ASD-EXP) (n=50); 2) children with ASD who will receive the intervention at the end of the trial (wait-list controls) (ASD-WLC) (n=50); 3) NT children with reading comprehension deficits who will receive intervention after their first MRI scan (NT-EXP) (n = 50); and 4) NT (n = 50) control participants (no reading comprehension deficits) who will be scanned twice but will not receive any intervention. A total of 200 participants (with 20 additional participants to account for attrition) will take part in this project. It should be noted that neuroimaging as well as behavioral studies of language in autism have largely ignored children with comprehension deficits. The proposed project addresses this critical gap by targeting brain plasticity in ASD and NT children (age: 7-13 years), with the following three independent, but inter-related specific aims.

AIM #1: Examine the differential impact of V/V intervention on the functional organization (activation and functional connectivity) of the brain's reading network (Koyama et al., 2011) in ASD and NT children who share reading comprehension deficits.

Hypothesis: Along with improvement in comprehension in both groups, the investigators predict that the connectivity between classic language areas and regions involved in visual/visuospatial processing will be stronger in ASD-EXP children compared to NT-EXP children after intervention.

AIM #2: Test the impact of V/V intervention on the microstructural connectivity of the white matter underlying reading network (primarily AF: the arcuate fasciculus and UF: the uncinate fasciculus) in ASD and NT children who share similar reading comprehension deficits.

Hypothesis: At post-scanning, white matter connectivity of the AF and UF (connecting frontal and temporal areas) will be increased in children who receive V/V intervention compared to themselves and to waitlist controls. It is expected that the extent of this change will differ between ASD-EXP and NT-EXP groups.

AIM #3: Establish brain-behavior relationship by testing how improvements in language skills (decoding, comprehension, fluency and other components) and autism symptoms predict post-intervention changes in neurobiological and behavioral profiles in ASD and NT children.

Hypotheses: 1) Improvement in comprehension (as measured by Gray Oral Reading Test) following V/V intervention will predict increased activation, functional connectivity, and white matter connectivity in the reading network in NT-EXP and ASD-EXP groups; 2) ASD symptom severity will negatively predict improvement in comprehension and in reading network response, and may help differentiate the nature of language deficits between ASD-EXP and NT-EXP groups.

The outcomes of this study will inform us about intervention-related changes in brain and behavior in ASD children with language deficits. This, in turn, may have translational significance in education. The inclusion of NT-EXP and NT control groups provide a unique opportunity to glean further into the nature of reading deficits in ASD and NT children and to the specificity of such deficits in ASD.

ELIGIBILITY:
Inclusion Criteria:

1. Full Scale and Verbal IQs > 70
2. be 7-13 years of age;
3. no antipsychotics for at least one month
4. no anti-epileptics/convulsants for at least one week
5. no stimulants for 24 hours prior to testing; and
6. subjects with ASD meet DSM-V criteria (American Psychiatric Association, 2013)
7. Neurotypical participants will be medically healthy (below ASD symptom cutoff score on the SCQ (Rutter, Bailey, & Lord, 2003); without a self-reported and parent- reported history of neurologic or psychiatric disorders; and without a family history of ASD)
8. The NT-EXP participants need to have similar profile of reading comprehension difficulties as the ASD participants with average decoding accompanied by below average reading comprehension.

Exclusion Criteria:

1. contraindication for MRI (cardiac pacemaker, aneurysm clip, cochlear implants, Intra Uterine Device, shrapnel, neurostimulators, defibrillator, artificial heart valve, or history of metal fragments in eyes, pregnancy, a body weight of more than 250 lbs. and claustrophobia)
2. seizure disorder or history of head injury

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2019-01-10 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Functional and anatomical changes in the brain | 10-12 weeks
  changes in the brain, measured by Magnetic Resonance Imaging, as a result of reading intervention
Change in reading comprehension | 10-12 weeks
  improvement in reading comprehension, measured by the Grey Oral Reading Test, as a result of reading intervention

SECONDARY OUTCOMES:
Relationship between neurobiological and behavioral changes | 10-12 weeks
  changes in reading comprehension, measured by GORT, will be related to the changes in brain organization (measured by MRI)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama, Tuscaloosa, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared through NIH Data Archive.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Data sharing through NDA has already been started; however, we have requested data to be made available to other researchers only after 2024.